CLINICAL TRIAL: NCT00470548
Title: Phase I/II Trial of Abraxane® (ABI-007) and Alimta® (Pemetrexed) in Advanced Solid Tumors With Emphasis on Non-Small Cell Lung Cancer (NSCLC) and Breast Cancer
Brief Title: Abraxane and Alimta in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Practice patterns with pemetrexed have evolved.
Sponsor: University of California, Davis (Other)
Collaborators: Celgene (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#185; 224355 (Other Grant/Funding Number: UC Davis); ABX027 (Other Grant/Funding Number: Celgene); H3E-US-I017 (Other Grant/Funding Number: Eli Lilly)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer; Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: male breast cancer; recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Breast Neoplasms, Male; Carcinoma, Non-Small-Cell Lung | interventions — Albumin-Bound Paclitaxel; Taxes; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I: Abraxane and Alimta (Experimental): Three dose levels were tested. Pemetrexed 500mg/m2 day 1 and nab-paclitaxel day 1 at 180, 220, and 260 mg/m2 every 21 days.
  Interventions: Drug: Abraxane; Drug: Alimta
- Phase II: Abraxane and Alimta (Experimental): Pemetrexed 500mg/m2 day 1 and nab-paclitaxel day 1 at 260 mg/m2 every 21 days.
  Interventions: Drug: Abraxane; Drug: Alimta

INTERVENTIONS:
Drug: Abraxane — ABI-007 IV administration following pemetrexed on Day 1 of each cycle (infused over 30 minutes)
  Other Names: paclitaxel albumin-stabilized nanoparticle formulation; ABI-007
Drug: Alimta — Pemetrexed IV administration on Day 1 of each cycle (infused over 10 minutes)
  Other Names: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving paclitaxel albumin-stabilized nanoparticle formulation together with pemetrexed may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of paclitaxel albumin-stabilized nanoparticle formulation when given together with pemetrexed and to see how well they work in treating patients with advanced non-small cell lung cancer, breast cancer, or other solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of paclitaxel albumin-stabilized nanoparticle formulation when administered with pemetrexed disodium in patients with advanced non-small cell lung cancer, breast cancer, or other solid tumors. (Phase I)
* Determine the efficacy of this regimen, as measured by objective tumor response rate (RECIST criteria), in these patients. (Phase II)

Secondary

* Determine the preliminary efficacy of paclitaxel albumin-stabilized nanoparticle formulation and pemetrexed disodium in these patients. (Phase I)
* Determine the overall survival of patients treated with this regimen. (Phase II)
* Evaluate the frequency and severity of toxicities associated with this regimen. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of paclitaxel albumin-stabilized nanoparticle formulation followed by an open-label, phase II study.

* Phase I: Patients receive pemetrexed disodium IV over 10 minutes and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of paclitaxel albumin-stabilized nanoparticle formulation until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive pemetrexed disodium and paclitaxel albumin-stabilized nanoparticle formulation at the MTD as in phase I.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria

1. For the phase II portion patients must have cytologically or histologically proven selected stage IIIB (pleural effusion) or IV NSCLC.
2. For the phase II portion patients must have NSCLC that has progressed or recurred after treatment with platinum-based therapy.
3. No prior pemetrexed. Prior Taxol is allowed. Prior ABI 007 is not allowed.
4. Patients must have measurable disease by RECIST criteria for the phase II portion.
5. Patients must be 18 years of age or older.
6. Patients must have a performance status of 0 -2
7. Patients must have an estimated survival of at least 3 months.
8. Any prior chemotherapy must have been completed at least 4 weeks prior to start of treatment.
9. Patients must have adequate renal function as documented by a calculated creatinine clearance of > 45 ml/min
10. Patients must have adequate liver functions: AST and ALT < 2.5 X upper limit of normal, and bilirubin < upper limit of normal.
11. Patients must have adequate bone marrow function: Platelets >100,000 cells/mm3 and ANC > 1,500 cells/mm3.
12. For patients who have baseline clinically significant pleural or peritoneal effusions (on the basis of symptoms or clinical examination) before initiation of pemetrexed therapy, consideration should be given to draining the effusion prior to dosing.
13. Patients with asymptomatic treated brain metastasis (surgical resection or radiotherapy) may be included if they are neurologically stable and have been off steroids and anticonvulsants for at least 4 weeks.
14. Patients must be able to take and retain oral medication.
15. Ability to take folic acid, vitamin B12 and dexamethasone according to protocol.
16. Ability to interrupt NSAIDS 2 days before, the day of, and 2 days following administration of pemetrexed.
17. Patients of reproductive potential must agree to use effective contraceptive method while on treatment and for 3 months afterwards as the effects of these drugs on the unborn fetus are unknown.
18. No other current active malignancy.
19. Patient or his/her legally authorized representative or guardian signed the Informed Consent form prior to participation in any study-related activities.

Exclusion Criteria

1. Pregnant or breastfeeding women.
2. Patient with pre-existing peripheral neuropathy of NCI CTCAE Version 3.0 of grade 2.
3. Patient has a clinically significant concurrent illness.
4. Patient is currently enrolled in a different clinical study in which investigational procedures are performed or investigational therapies are administered.
5. Patient has a history of allergy or hypersensitivity to the study drugs or a taxane.
6. Patient has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug.
7. Prior therapy with pemetrexed, or ABI-007.
8. Patient is receiving treatment with any excluded concomitant medication.
9. Presence of third space fluid which cannot be controlled by drainage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Gandara, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

REFERENCES:
- [Result] Ho C, Davies AM, Sangha RS, Lau D, Lara P Jr, Chew HK, Beckett L, Mack PC, Riess JW, Gandara DR. Phase I/II trial of pemetrexed plus nab-paclitaxel in advanced solid tumor patients with emphasis on non-small cell lung cancer. Invest New Drugs. 2013 Dec;31(6):1587-91. doi: 10.1007/s10637-013-0024-y. Epub 2013 Sep 8. PMID 24013936

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Level 1: Pemetrexed 500 mg/m2 plus Abraxane 180 mg/m2
- Phase I: Dose Level 2: Pemetrexed 500 mg/m2 plus Abraxane 220 mg/m2
- Phase I: Dose Level 3; Phase II: Pemetrexed 500 mg/m2 plus Abraxane 260 mg/m2
Period: Overall Study
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase I: Dose Level 3 | Phase II
Started | 3 | 3 | 6 | 37
Completed | 3 | 3 | 6 | 37
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Abraxane and Pemetrexed: A 3 + 3 dose escalation design was used to determine the maximum tolerated dose and the recommended phase II dose. Alimta® (pemetrexed) 500 mg/m2 IV administration on Day 1 of each cycle with Abraxane® (ABI 007) 180 mg/m2, 220 mg/m2 and 260 mg/m2 IV administration following pemetrexed on Day 1 of each cycle .
- Phase II: Abraxane and Pemetrexed: Alimta® (pemetrexed) 500 mg/m2 IV administration on Day 1 of each cycle with Abraxane® (ABI 007) 260 mg/m2IV administration following pemetrexed on Day 1 of each cycle
- Total: Total of all reporting groups
Arm/Group | Phase I: Abraxane and Pemetrexed | Phase II: Abraxane and Pemetrexed | Total
Number analyzed (Participants) | 12 | 37 | 49
Age, Continuous [Median (Full Range); unit: years] | 70 [51 to 76] | 63 [45 to 77] | 63 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 19
  Male | 7 | 23 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 37 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Dose limiting toxicity (DLT) was defined as any of the following occurring during the first cycle: Grade 4 thrombocytopenia, or grade 3 thrombocytopenia associated with bleeding, requirement for transfusion, febrile neutropenia, neutropenia with documented infection. Non-hematologic DLT included any other ≥ grade 3 non-hematologic toxicity that was clinically significant and considered by the investigator to be related to study drug. Alopecia and grade 3 allergic reaction/hypersensitivity with infusion were not considered DLTs.
Time Frame: Up to21 days
Population: At dose level 1, 2 and 3 three participants were treated with no dose limiting toxicities. Three additional participants were treated at dose level 3 with no dose limiting toxicities.
Measure: Number; unit: participants
Groups:
- Phase I: Dose Level 1: A 3 + 3 dose escalation design was used to determine the maximum tolerated dose and the recommended phase II dose. Alimta® (pemetrexed) 500 mg/m2 IV administration on Day 1 of each cycle with Abraxane® (ABI 007) 180 mg/m2 IV administration following pemetrexed on Day 1 of each cycle .
- Phase I: Dose Level 2: A 3 + 3 dose escalation design was used to determine the maximum tolerated dose and the recommended phase II dose. Alimta® (pemetrexed) 500 mg/m2 IV administration on Day 1 of each cycle with Abraxane® (ABI 007) 220 mg/m2 IV administration following pemetrexed on Day 1 of each cycle .
- Phase I: Dose Level 3: A 3 + 3 dose escalation design was used to determine the maximum tolerated dose and the recommended phase II dose. Alimta® (pemetrexed) 500 mg/m2 IV administration on Day 1 of each cycle with Abraxane® (ABI 007) 260 mg/m2 IV administration following pemetrexed on Day 1 of each cycle .
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase I: Dose Level 3
Number analyzed (Participants) | 3 | 3 | 6
participants | 0 | 0 | 0

2. Primary Outcome: Number of Patients With Toxicities
Description: Toxicities was evaluated based on the standard NCI CTCAE Version 3.0 grading criteria. Attributable grade ≥ 3 hematologic and non-hematologic toxicities are presented here.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: Pemetrexed and Abraxane: Pemetrexed 500 mg/m2 plus Abraxane 260 mg/m2
Arm/Group | Phase II: Pemetrexed and Abraxane
Number analyzed (Participants) | 37
Participants | 15

3. Secondary Outcome: Duration of Overall Survival
Description: From time of enrollment to the first observation of disease progression or death.
Time Frame: Up to 2 years
Population: Of the 12 patients in the phase I component 10 were assessable for response. In the phase II component, 31 of 37 patients were evaluable for response.
Measure: Median (Standard Error); unit: months
Arm/Group | Phase I: Abraxane and Pemetrexed | Phase II: Abraxane and Pemetrexed
Number analyzed (Participants) | 10 | 31
months | 13.5 (0) | 4.5 (0)

4. Secondary Outcome: Number of Participants With Complete Response
Description: Per RECIST criteria, complete response (CR) is defined as the disappearance of all target lesions.
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Phase I: Abraxane and Pemetrexed | Phase II: Abraxane and Pemetrexed
Number analyzed (Participants) | 12 | 37
participants | 0 | 0

5. Secondary Outcome: Number of Participants With Stable Disease
Description: Stable Disease is measured from the start of the treatment until the criteria for disease progression are met. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Abraxane and Pemetrexed | Phase II: Abraxane and Pemetrexed
Number analyzed (Participants) | 12 | 37
Participants | 7 | 12

6. Secondary Outcome: Number of Participants With Partial Response
Description: At least a 30% decrease in the sum of the longest diameter of target lesions
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Abraxane and Pemetrexed | Phase II: Abraxane and Pemetrexed
Number analyzed (Participants) | 12 | 37
Participants | 0 | 5

7. Secondary Outcome: Number of Participants With Disease Control
Description: Disease control is complete response plus partial response plus stable disease from the start of treatment to death or disease progression.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Abraxane and Pemetrexed | Phase II: Abraxane and Pemetrexed
Number analyzed (Participants) | 12 | 37
Participants | 7 | 17

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Adverse events until they are resolved or stabilized, the patient is lost to follow-up, or the event is otherwise explained.
Arm/Group | Phase I: Abraxane and Alimta | Phase II: Abraxane and Alimta
Serious Adverse Events (participants affected / at risk) | 1/12 | 6/37
Other Adverse Events (participants affected / at risk) | 8/12 | 15/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Abraxane and Alimta (N=12) | Phase II: Abraxane and Alimta (N=37)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Fever (General disorders) | 0 | 1
Cardiac Ischemia (Cardiac disorders) | 0 | 1
Nasal Hemorrhage (Blood and lymphatic system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Skin Infection (Infections and infestations) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Abraxane and Alimta (N=12) | Phase II: Abraxane and Alimta (N=37)
Anemia (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Cardiac Ischemia (Cardiac disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Hypersensitivity (General disorders) | 0 | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 | 1
Increased transaminases (Blood and lymphatic system disorders) | 0 | 1
Sensory neuropathy (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The phase II portion accrued 37 patients before early closure due to increasing the first-line pemetrexed/platinum doublet use in non-squamous NSCLC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes